CLINICAL TRIAL: NCT00005748
Title: Stress Reduction and Prevention of Hypertension in Blacks
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5056; R01HL060703 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2005-03

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

SUMMARY:
To examine the role of Transcendental Meditation in stress reduction and prevention of hypertension in Blacks.

DETAILED DESCRIPTION:
BACKGROUND:

African Americans suffer from disproportionate rates of hypertension and related cardiovascular morbidity and mortality due, at least in part, to excessive socioenvironmental and psychosocial stress. Furthermore, despite the substantial individual and population risk burden associated with high normal blood pressure (BP) in African Americans, there had been no controlled studies to evaluate stress reduction approaches in the primary prevention of hypertension targeted to this high risk group. Therefore, recent (mid 1990s) NIH and NIMH policy committees called for a new research focus on primary prevention of hypertension targeted to high risk populations-notably African Americans with high normal BP. In previous randomized controlled trials by the investigator, hypertension and psychosocial stress were significantly reduced in low SES African Americans who practiced stress reduction with the Transcendental Mediation (TM) program compared to relaxation or health education controls. In the most recent long-term trial, African Americans with borderline hypertension showed BP reductions that would be associated with a 17 percent decrease in prevalence of hypertension, a 15 percent reduction in stroke, and a 6 percent reduction in CHD in the population. These BP reductions compared favorably to decreases shown with sodium restriction and weight loss programs in other prevention trials. Also, pilot data from two clinical trials indicated that TM was associated with significantly lower cardiovascular morbidity and mortality in African Americans and in Caucasians with high BP over a 5-year and 15-year period, respectively.

DESIGN NARRATIVE:

A randomized controlled trial of stress reduction for the primary prevention of hypertension was conducted in African Americans with high normal BP. African American males and females (N-352, aged 21-75 years) with high normal BP (SBP 130-139 and/or DBP 85-89 mm Hg) were recruited from the African American Family Heart Health Plan at the Medical College of Wisconsin, Milwaukee, which housed the nation's largest registry of African Americans with known CVD risk factors. After baseline assessment, participants were randomized to either the TM program or to a matched health education control intervention. The primary outcome was change in clinic BP over a 12-month follow-up. Secondary outcomes included changes in ambulatory BP, hypertensive events, psychosocial stress and health behaviors. Also, a model of the pathways through which components of stressful experience affect high BP in African Americans was tested.

This study is described as a clinical trial. The summary statement states that it is not an NIH Phase III clinical trial.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-05; Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Schneider — Maharishi University